CLINICAL TRIAL: NCT05315843
Title: Cobalamin Supply and Metabolism in Healthy Children From Birth to the Age of 12 Months and in Their Mothers (Cbl_Neo)
Acronym: Cbl_Neo
Status: Completed | Type: Observational
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: Cbl_Neo
Record Dates: First submitted 2022-03-31; First posted 2022-04-07 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Vitamin B 12 Deficiency
MeSH Terms: conditions — Vitamin B 12 Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Introduction: Infants with severe vitamin B12 (cobalamin, Cbl) deficiency can develop severe, sometimes irreparable neurological damage in the first months of life. Neonatal Cbl deficiency is usually secondary and due to low maternal Cbl stores, e.g. in vegan diets or pernicious anaemia. This Cbl deficiency is then often also found in breast milk. In the Austrian newborn screening (NBS) for congenital diseases of the Cbl metabolism, newborns with secondary Cbl deficiency are also frequently discovered. For these, the risk-benefit assessment of the invasive work-up and treatment that follows is complex. Little is known about how Cbl levels in maternal blood relate to those in breast milk and the corresponding levels in the child.

Objective: To investigate the effects of maternal nutrition and maternal Cbl status on neonatal Cbl levels. In the breastfeeding period, the effects of maternal nutrition on breast milk and infant Cbl status will be investigated, as well as their relationship to the maternal and infant microbiome. We hypothesise that adequate Cbl supply in early life is not determined by diet alone, but also by the interactions between diet and microbiome.

Design and methods: Prospective cohort studies of 100 women and their children with measurement of Cbl, methylmalonic acid, homocysteine and other metabolites of Cbl metabolism in umbilical cord blood, maternal blood, dried blood spots and urine from the child at birth. The same parameters are measured in the mother's blood and breast milk after 3 and 9 months; in the child, only measurements of methylmalonic acid in the urine are carried out. A 3-day dietary record is taken from the mother at all measurement times, and from the child at the measurement times of 3 and 9 months. Stool is collected from mother and child at all measurement time points to examine the microbiome relevant to Cbl metabolism. A child development interview will be conducted with mothers by telephone at 12 months of age of their child.

Schedule: The study lasts 2 years with pre- and post-processing. The LKH Bregenz has about 1200 births per year. Assuming a willingness to participate in the study and an enrolment rate of about 20% of the women, a recruitment period of 6 months is planned (enrolment of first participant day 1, last participant end of study month 6; last laboratory parameter measurement end of study month 15; last child development interview study month 18).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* their newborns

Exclusion Criteria:

* children: preterm birth
* children: neonatal disease
* women: disease around birth
* women: multiples pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant females and their children
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Homocysteine | 9 months
  Plasma total Homocysteine higher in B12 deficient children

CONTACTS AND LOCATIONS:
Locations (2):
- LKH Bregenz, Bregenz, Austria
- University Childrens Hospital Freiburg, Freiburg im Breisgau, Germany

IPD SHARING:
Plan to Share IPD: No